CLINICAL TRIAL: NCT06110598
Title: CAPEcitabine eXtension of Adjuvant Therapy for Pancreatic Adenocarcinoma: (CAPE-X)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3223
Record Dates: First submitted 2023-10-19; First posted 2023-10-31 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Pancreas Cancer; Pancreas Adenocarcinoma
Keywords: pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to the treatment arm. There will be no blinding of participants and the trial will not be placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Extended adjuvant therapy with capecitabine (Experimental): * Participants randomized to Arm A will take capecitabine (1000mg by mouth twice a day, 3-week cycle [2 weeks on therapy, 1 week off]) for up to 18 cycles, or until progression or intolerance to therapy develops.
  * Participants who remain without disease recurrence at completion of 18 cycles of therapy who wish to continue therapy may do so at the discretion of their treating medical oncologist. Participants will be followed at standard 12-week intervals, where they will undergo routine cross-sectional imaging and labs.
  Interventions: Drug: Capecitabine
- Arm B: Active surveillance (No Intervention): * Participants randomized to Arm B will undergo active surveillance, with no active treatment for the duration of their participation in the study.
  * Participants in Arm B will undergo re-staging every 12 weeks (+/- 7 days), consisting of cross-sectional imaging (CT or PET-CT) and labs (CBC, chemistry panel, CA19-9 and blood draw for ctDNA). In addition to re-staging every 12 weeks, participants may be seen by their medical or surgical oncologist as clinically indicated. Participants who experience disease relapse may transition to palliative systemic therapy or best supportive care at the discretion of their treating medical oncologist.

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is an oral prodrug that is enzymatically converted to 5-fluorouracil (5-FU) in vivo. Both normal and tumor cells metabolize 5-FU to 5-fluoro-2'-deoxyuridine monophosphate (FdUMP) and 5-fluorouridine triphosphate (FUTP). These metabolites cause cell injury by two different mechanisms. First, FdUMP and the folate cofactor, N5-10-methylenetetrahydrofolate, bind to thymidylate synthase (TS) to form a covalently bound ternary complex. This binding inhibits the formation of thymidylate from 2'-deoxyuridylate. Thymidylate is the necessary precursor of thymidine triphosphate, which is essential for the synthesis of DNA, so that a deficiency of this compound can inhibit cell division. Second, nuclear transcriptional enzymes can mistakenly incorporate FUTP in place of uridine triphosphate (UTP) during the synthesis of RNA. This metabolic error can interfere with RNA processing and protein synthesis.
  Other Names: Xeloda®
  Arms: Arm A: Extended adjuvant therapy with capecitabine

SUMMARY:
* This study is being done to find out if extending adjuvant chemotherapy for patients by giving additional chemotherapy can lengthen the amount of time before their cancer comes back. The additional chemotherapy is called capecitabine.
* Capecitabine is an oral drug (taken by mouth). It is approved by the US Food and Drug Administration (FDA) for adjuvant treatment of adults with pancreatic cancer and also for the treatment of other types of cancer

DETAILED DESCRIPTION:
- Pancreatic adenocarcinoma remains one of the deadliest common solid tumor malignancies with an overall survival of 11% at 5 years for all comers. Approximately 50% of patients present with metastatic disease at the time of diagnosis. Approximately 20% of patients have localized disease at diagnosis and are candidates for surgical resection, which is necessary but not sufficient for long-term survival, and the most optimal survival outcomes are seen with multimodal therapy. The recently published SWOG S1505 study demonstrated that participants with localized pancreatic adenocarcinoma treated with either of the two most active multi-agent regimens (FOLFIRINOX or gemcitabine with nab-paclitaxel) in the perioperative setting had a median recurrence-free survival of 10.9-14.2 months, and 2-year overall survival of 47-48% (median: 23.2 vs. 23.6 months), which is similar to outcomes observed in older studies examining the efficacy of gemcitabine monotherapy or 5-FU monotherapy.

Currently, there are no guideline recommendations for extension of adjuvant therapy upon completion of all standard therapy (defined as surgery, multi-agent chemotherapy, + radiotherapy) for localized pancreatic adenocarcinoma. EA2192 (APOLLO; https:// clinicaltrials. gov/ct2/show/NCT04858334), a phase II randomized controlled trial, is currently accruing and investigating the efficacy of twelve months of olaparib on relapse-free survival in participants with germline BRCA- or PALB2-mutated pancreatic adenocarcinoma, which accounts for a small minority (4-7%) of cases. Olaparib was found to improve progression-free survival in participants with germline-mutated BRCA or PALB2 metastatic pancreatic adenocarcinoma. There are no trials examining extension of adjuvant therapy after completion of all standard therapy in the non-genomically selected patients with localized disease, who comprise 93-96% of these pancreas cancer patients.

- This study will be a phase 2 randomized clinical trial, with a 2:1 merged blocked, stratified randomization to the treatment arm to test the efficacy of extended adjuvant therapy in delaying disease relapse following completion of all standard therapy for localized pancreatic adenocarcinoma, as compared to the standard of care, which is active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed pancreatic adenocarcinoma.
* Participants must have undergone curative-intent surgical resection and received at least 4 months of multi-agent cytotoxic chemotherapy, regardless of treatment sequence or chemotherapy backbone.
* Participants must be within 12 weeks of completion of standard perioperative therapy (defined as resection, multi-agent systemic chemotherapy, + radiotherapy, regardless of treatment sequence).
* Participants must have absence of or unknown BRCA1, BRCA2, or PALB2 germline or somatic mutational status.
* Participants must have no evidence of recurrent disease.
* Age >18 years because no high-quality dosing or adverse event data are currently available on the use of capecitabine in in participants ≤18 years of age. Additionally, pancreatic adenocarcinoma is exceedingly rare in participants <18 years of age. Therefore, children are excluded from this study.
* ECOG(Eastern Cooperative Oncology Group) Performance status < 2.
* Participants must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 10.0 g/dl
  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST(Aspartate aminotransferase) (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine within normal institutional limits
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment toxicities resolved to ≤ Grade 3 according to NCI CTCAE Version 5.0 (list exceptions, e.g. alopecia, neuropathy, fatigue, etc).
* Participants receiving any other investigational agents or participating in clinical trials that use OS or PFS(progression-free survival) as their primary or secondary endpoints would prohibit participation in the current study. Patients enrolled or previously enrolled in non-therapeutic trials, or trials with only correlative endpoints are allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine or 5-fluorouracil.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with known low or absent dihydropyimidine dehydrogenase (DPD)activity
* Women who are pregnant or breastfeeding are excluded from this study because capecitabine is a category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with capecitabine, breastfeeding should be discontinued if the mother is treated with capecitabine.
* Participants who are known to be HIV-positive on combination antiviral therapy are ineligible because of the potential for pharmacokinetic interaction with capecitabine. In addition, these participants are at increased risk of lethal infections when treated with marrow suppressive therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | Assessed every 3 months from the date of randomization until the first documentation of disease relapse or death, up to 24 months, and then every 6 months after the initial 24 months up to 4 years
  Relapse-free survival (RFS), defined as the time from randomization to first documentation of disease relapse or death, defined as radiographic evidence of local or distant primary tumor relapse, whichever occurs first; participants alive without relapse will be censored at the date of last disease assessment.

SECONDARY OUTCOMES:
Overall survival (OS) | Assessed every 3 months from the date of randomization until the first documentation of disease relapse or death, up to 24 months, and then every 6 months after the initial 24 months up to 4 years
  Overall survival (OS), defined as the time from randomization to death from any cause; participants still living will be censored at the date last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Ocuin, MD, FACS, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals, Cleveland Medical Center, Seidman Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underline results reported in this publication after deidentification
Supporting Information: Study Protocol
Time Frame: Starting 9 months and ending 36 months following article publication